CLINICAL TRIAL: NCT05222841
Title: The Effectiveness of the Spermotrend Food Supplement in the Treatment of Male Infertility and Benign Prostatic Hyperplasia
Brief Title: The Effectiveness of Spermotrend Food Supplement in the Treatment of Male Infertility
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPT-NICA-2021
Record Dates: First submitted 2021-10-18; First posted 2022-02-03 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-01

CONDITIONS: Male Infertility; Benign Prostatic Hyperplasia; Spermatogenesis and Semen Disorders
Keywords: Antioxidant; spermatogenesis; Male infertility; Benign Prostatic Hyperplasia; Pygeum africanum
MeSH Terms: conditions — Infertility, Male; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spermotrend (Experimental)
  Interventions: Dietary Supplement: Spermotrend

INTERVENTIONS:
Dietary Supplement: Spermotrend — Patients who are treated with Spermotrend (536,62g) are given 3 capsules every day for 3 months, taken orally every 8 hours.

SUMMARY:
Spermotrend is a natural based product manufactured by Catalysis Laboratories. Its composition contains different essential elements for spermatogenesis: selenium, zinc and fructose. In addition, it contains L-arginine, natural precursor of nitric oxide that favors vasodilation, and pygeum africanum extract with antioxidant, antiinflammatory, antiandrogenic and antiproliferative action.

Its main action resides in the control of oxidative damage to the tissues of the male reproductive system, as well as the control of correct spermatogenesis.

Given that sperm quality can be altered by oxidative stress and that male infertility affects more and more people, the prevention and management of this deterioration becomes increasingly important.

Therefore, to evaluate Spermotrend as a new therapy for male infertility, the investigators are going to study the safety and efficacy of this treatment in this clinical trial.

RESEARCH HYPOTHESIS

The treatment with Spermotrend improves the parameters of the spermatogenesis.

GENERAL OBJECTIVES

To evaluate the effectiveness and the safety level of the natural Spermotrend product in the treatment of male infertility.

SPECIFIC OBJECTIVES

* Evaluate the increase in sperm motility and concentration.
* Identify the improvement in the seminal fluid volume.
* Identify the positive changes in the sperm morphology.
* Determine how to maintain the semen analysis in a normal range.
* Describe the adverse effects.

SECONDARY OBJECTIVES

* Identify the improvement in urinary symptoms related with benign prostatic hyperplasia.
* Identify the improvement in varicocele.

DETAILED DESCRIPTION:
Every day, all over the world, increasingly more couples have to go to specialised centres in the hope of solving their infertility problems. In the past, female infertility was thought to be the main cause of this problem, but in the course of time, those of us who work in the field of Gynaecology, which is such a delicate issue, are convinced that the initial statistics concerning the prevalence of infertility in women is now just pure myth. The male factor is the main cause of infertility in numerous couples that go to the doctor every day, the percentage of which surpasses that of female infertility in many places. Not everyone have access to the high-tech assisted reproduction techniques which compensate for any spermatogenesis. Many studies have been carried out in the hope of improving the sperm quality in men. Antioxidants play an important role in the spermiogenesis, but so far no product has been found that really meets the expectations of improving the spermatogenesis in the short term. A product that naturally or through low- tech assisted reproduction techniques improves the pregnancy rates among couples that suffer from this type of disorder.

Catalysis Laboratories is specialized in natural antioxidant products as adjuvants and alternative treatments for prevention, management and recovery from different diseases.

The aim of this clinical trial is to study the efficacy and safety of Spermotrnend, a natural product manufactured by Catalysis Laboratories, in the improvement of sperm's quality and quantity in male infertility as well as in urinary symptoms and varicocele in those patients who suffer it in association or not with infertility.

ELIGIBILITY:
Inclusion Criteria:

* Males over 18.
* Patient who shows alterations of the spermatogenesis and/or benign prostatic hyperplasia.
* Patients without testicular pathology.
* Serology and HIV negative.
* Signed informed consent.

Exclusion Criteria:

* Patients with associated pathologies: epididymo-orchitis, radiation or chemotherapy.
* Patients with a testicular pathology that has been resolved.
* Patients with non-transmissible chronic pathologies.
* Patients who have not agreed to take part in the study.
* Patients that are undergoing antioxidant treatment or who have completed this treatment in the last six months.
* Patients who are being treated with vitamins or who have completed this treatment in the last six months.
* Patients that are being treated with anti-inflammatory medications or who have completed this treatment in the last six months.
* Patients who are undergoing hormone treatment prescribed for andrology or who have completed this treatment in the last six months.
* Patients with serology or who are HIV positive.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Sperm motility | 3 months
  Evaluate the change in sperm motility by spermiogram.
Sperm concentration | 3 months
  Evaluate the changes in sperm concentration by spermiogram.
Seminal fluid volume. | 3 months
  To identify the changes in the seminal fluid volume by spermiogram.
Sperm morphology. | 3 months
  Identify the changes in the sperm morphology by spermiogram.
Incidence of adverse events during the treatment with Spermotrend | 3 months
  To study and asses any adverse event related with the product assay in patients with male infertility, measured by means of a bimonthly personal questionnaire: nausea, vomiting, digestive pain, stomach ache... (mild, moderate, severe, yes or no).

SECONDARY OUTCOMES:
Maintenance of semen quality in a normal range. | 6 months
  Time of maintenance of the semen quality spermiogram analysis compared to the base line (weeks/months).
Evaluation of the function of the urinary bladder and urethra | 3 months
  Residual urine will be determined by urodynamic evaluation (Volume in mL).
Evaluation of the function of the urinary bladder and urethra | 3 months
  Urine flow rates (Qmax) will be determined by urodynamic evaluation (milliliters).
Clinical evoluation of Benign prostatic hyperplasia | 3 months
  To evaluate the urinary symptoms related with benign prostatic hyperplasia by blood analysis: AUA guideline prostate-specific antigen (PSA) and serum creatinine measurements will be measured to evaluate the benign prostatic hyperplasia . Serum PSA level should be determined in men in the BPH age group, preferably before the rectal examination. A careful history taking and physical examination will usually identify patients at risk for bleeding tendencies.
Evaluation of urinary symptoms related with benign prostatic hyperplasia | 3 months
  To evaluate the urinary symptoms related with benign prostatic hyperplasia by the specific questionnaire International Prostate Symptom Score (IPSS). Answers will be scored from 0=Not at all; 1= Less than 1 time in 5; 2=Less than half of time; 3= About Half of time; 4=More than half of time; to 5= Almost always.
  (For example: - How often have you haf the sensation of not emptying your bladder completely after you finished urinating? From 0 to 5).
  The summatory of symptom scores will be evaluated as 1-7 mild symptoms; 8-19 moderate symptoms; and 20-35 severe symptoms.
Prostate size in patients with benign prostatic hyperplasia | 3 months
  To evaluate the benign prostatic hyperplasia volume by image analysis with ultrasound. Residual urine and urine flow rates will be determined by urodynamic evaluation.
Varicocele Degree | 3 months
  To evaluate varicocele degree (1, 2 or 3) in term of size and its evolution in male infertility from the base line to the end of the treatment with Spermotrend.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Seniors Managua, Managua, Nicaragua

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Boitani C, Puglisi R. Selenium, a key element in spermatogenesis and male fertility. Adv Exp Med Biol. 2008;636:65-73. doi: 10.1007/978-0-387-09597-4_4. PMID 19856162
- [Background] H B, A S, A J, P A, B S, D S, A EM, M N. Radioprotective Effects of Zinc and Selenium on Mice Spermatogenesis. J Biomed Phys Eng. 2020 Dec 1;10(6):707-712. doi: 10.31661/jbpe.v0i0.957. eCollection 2020 Dec. PMID 33364208
- [Background] Naderi M, Ahangar N, Badakhshan F, Ghasemi M, Shaki F. Zinc and selenium supplement mitigated valproic acid-induced testis toxicity by modulating the oxidative redox balance in male rats. Anat Cell Biol. 2021 Sep 30;54(3):387-394. doi: 10.5115/acb.20.280. PMID 34588319
- [Background] Irani M, Amirian M, Sadeghi R, Lez JL, Latifnejad Roudsari R. The Effect of Folate and Folate Plus Zinc Supplementation on Endocrine Parameters and Sperm Characteristics in Sub-Fertile Men: A Systematic Review and Meta-Analysis. Urol J. 2017 Aug 29;14(5):4069-4078. PMID 28853101
- [Background] Kerns K, Zigo M, Sutovsky P. Zinc: A Necessary Ion for Mammalian Sperm Fertilization Competency. Int J Mol Sci. 2018 Dec 18;19(12):4097. doi: 10.3390/ijms19124097. PMID 30567310
- [Background] Allouche-Fitoussi D, Breitbart H. The Role of Zinc in Male Fertility. Int J Mol Sci. 2020 Oct 21;21(20):7796. doi: 10.3390/ijms21207796. PMID 33096823
- [Background] Madej D, Pietruszka B, Kaluza J. The effect of iron and/or zinc diet supplementation and termination of this practice on the antioxidant status of the reproductive tissues and sperm viability in rats. J Trace Elem Med Biol. 2021 Mar;64:126689. doi: 10.1016/j.jtemb.2020.126689. Epub 2020 Nov 19. PMID 33248336
- [Background] Cicero AFG, Allkanjari O, Busetto GM, Cai T, Largana G, Magri V, Perletti G, Robustelli Della Cuna FS, Russo GI, Stamatiou K, Trinchieri A, Vitalone A. Nutraceutical treatment and prevention of benign prostatic hyperplasia and prostate cancer. Arch Ital Urol Androl. 2019 Oct 2;91(3). doi: 10.4081/aiua.2019.3.139. PMID 31577095
- [Background] Santos HO, Howell S, Teixeira FJ. Beyond tribulus (Tribulus terrestris L.): The effects of phytotherapics on testosterone, sperm and prostate parameters. J Ethnopharmacol. 2019 May 10;235:392-405. doi: 10.1016/j.jep.2019.02.033. Epub 2019 Feb 18. PMID 30790614
- [Background] Salinas-Casado J, Esteban-Fuertes M, Carballido-Rodriguez J, Cozar-Olmo JM. Review of the experience and evidence of Pygeum africanum in urological practice. Actas Urol Esp (Engl Ed). 2020 Jan-Feb;44(1):9-13. doi: 10.1016/j.acuro.2019.08.002. Epub 2019 Oct 16. English, Spanish. PMID 31627963
- [Background] Shenouda NS, Sakla MS, Newton LG, Besch-Williford C, Greenberg NM, MacDonald RS, Lubahn DB. Phytosterol Pygeum africanum regulates prostate cancer in vitro and in vivo. Endocrine. 2007 Feb;31(1):72-81. doi: 10.1007/s12020-007-0014-y. PMID 17709901
- [Background] Pagano E, Laudato M, Griffo M, Capasso R. Phytotherapy of benign prostatic hyperplasia. A minireview. Phytother Res. 2014 Jul;28(7):949-55. doi: 10.1002/ptr.5084. PMID 25165780
- [Background] Larre S, Camparo P, Comperat E, Boulbes D, Haddoum M, Baulande S, Soularue P, Costa P, Cussenot O. Biological effect of human serum collected before and after oral intake of Pygeum africanum on various benign prostate cell cultures. Asian J Androl. 2012 May;14(3):499-504. doi: 10.1038/aja.2011.132. Epub 2011 Dec 26. PMID 22198631